CLINICAL TRIAL: NCT02873000
Title: A Prospective Randomized Trial of Incentive Spirometry in Non-critically Ill Hospitalized Patients With Shortness of Breath
Brief Title: Incentive Spirometry in Non-critically Ill Hospitalized Patients With Acute Respiratory Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jewish Hospital, Cincinnati, Ohio (Other)
Responsible Party: Principal Investigator, Imran Naqvi, Chief Hospitalist, Associated Program Director, Jewish Hospital, Cincinnati, Ohio
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-20
Record Dates: First submitted 2015-11-20; First posted 2016-08-19 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Pulmonary Complication; Dyspnea; Pneumonia; COPD; CHF; Atelectasis; PE
Keywords: incentive spirometry; outcome; length of stay,; hospital complication; general internal medicine; hospital medicine; non-critically-ill
MeSH Terms: conditions — Dyspnea; Pneumonia; Pulmonary Disease, Chronic Obstructive; Pulmonary Atelectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine Care Group (No Intervention): Routine Care (R): Standard of care therapy based on admitting diagnosis
- Experimental Group (Experimental): Intervention 1 (E1): addition of incentive spirometry every hour while awake;
  There will be a computerized protocol with specific instructions documenting:
  1. compliance
  2. patient position while using [sitting up vs laying flat in bed]
  3. inspiratory volume attained
  4. effort, motivation and compliance will subjectively be documented using a visual analogue 0-5 point scale.
  Interventions: Behavioral: Incentive Spirometry

INTERVENTIONS:
Behavioral: Incentive Spirometry — Incentive Spirometer is a tool that allows for deep breathing in a controlled setting while providing the user with visual feedback demonstrating the inspiratory volume of each breath.
  Arms: Experimental Group

SUMMARY:
To evaluate the use of Incentive Spirometry in Non-critically Ill Hospitalized Patients With Shortness of Breath.

DETAILED DESCRIPTION:
In recent years the focus in medicine has shifted towards efficient utilization of resources and improving patient outcomes. Incentive spirometry (IS) is a tool that mimics the natural process of yawning or sighing by allowing the user to take deep breaths in a controlled setting. This is a lung inflating maneuver that has been suggested to decrease the rate of pulmonary complications. The focus of utilization of IS and current studies has been predominantly on the post-operative surgical patient population. The mechanism of pulmonary complications in surgical patients is mixed in etiology possibly related to anesthesia, analgesics, pain and immobility leading to shallow breathing and subsequent atelectasis with concurrent hypoxia and risk of infection. The use of lung expanding maneuvers such as that provided by IS are thought to counteract shallow breathing thereby improving pulmonary outcomes. However, contrary to physiological theory, multiple studies and meta-analysis have failed to demonstrate its efficacy. The results of these studies are in direct conflict with what is expected scientifically.

The authors of this paper set out to find the reason for discordant data in existing literature, and found that there have been multiple methodological limitations associated with existing studies; hence, interpretation and recommendations based on current data should be done with caution. The common denominator in repeated criticisms of existing studies is lack of reporting on patient compliance with IS after it is prescribed. This is a major confounder, in clinical experience IS is often observed sitting dormant at patients' bedside. These observations are in synchrony with criticisms reported in literature and raise serious questions about validity of existing data that should be acknowledged. Despite lack of convincing evidence, IS is routinely prescribed by physicians in hospital medicine. IS is a low cost tool, nevertheless, the increasing frequency of its use is accumulating to a larger proportion of health care costs. This calls for further evaluation with a study of higher methodological quality to address the limitations of prior studies.

The scope of this study is different than that of existing studies in that it will evaluate the utility of IS in general medical patients. The sub-set of patients that are the focus of this study are those admitted with the chief complaint of "shortness of breath." The disease process in the former group leading to shortness of breath includes fluid over-load such as that in congestive heart failure, or an underlying lung process such as pneumonia, COPD, and/or pulmonary embolism. There is a parallel between mechanism of hypoxia in these patients and surgical patients in that these patients too often have pain and take high doses of analgesics, have shallow monotonous breathing and are immobile for long periods of time. From a physiological standpoint sustained maximal inhalation maneuvers may reverse and prevent progression of atelectasis by maintaining airway patency in all patients with shallow breathing of varying etiology not just the surgical sub-set.

In a tertiary center community teaching hospital the effectiveness of IS in general medical wards will be evaluated using a single center randomized clinical trial. The goal is to offer a study that overcomes the limitations of prior studies. Lack of strong evidence based data has led to inconsistencies in practice of physicians leading to higher health care costs. The authors hope to design a study of high methodological quality to assess the effectiveness of IS in medical patients; thereby closing the knowledge gap in evidence based practices that may aid physicians in their decision to utilize IS.

ELIGIBILITY:
Inclusion:

* Patients presenting to the ED with chief complaint of "shortness of breath," admitted to the hospitalist service
* Age >65 yrs of age

Exclusion:

* Patients who can not follow instructions/use IS device
* Cognitive impairment (Dementia/delirium/Developmental delay)
* Heavy sedation
* Inability to take part in deep breathing due to pain or diaphragmatic dysfunction
* Suicide or psych watch
* Patients under isolation
* ICU admission or care within the last 48 hours
* Recent hospitalization 30 days.
* Intubation within the last 60 days
* Routine care group patients that have IS prescribed to them by the admitting MD
* Chronic/Home oxygen dependence

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-04 (Estimated); Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Change in Forced Vital Capacity (FVC) | From admission to the hospital up to 48 hours
  FVC will be measured on admission and at 48 hours

SECONDARY OUTCOMES:
Subjective perception of respiratory distress | From admission to the hospital up to 48 hours
  Visual analogue scale (score 0-5) will be used to measure patient's subjective perception of respiratory distress on the day of admission, at 24 hours and at 48 hours.
Length of Stay (LOS) | Starting on admission and until discharge from the hospital (up to 14 days)
  Actual length of stay measured in days from date of admission to discharge will be reported per subject per group.
Pulmonary complications | Starting on admission and continuing for 7 days
  The total number of complications will be reported for each subject: i) radiographically as defined by the radiologist as new or worsening: atelectasis/consolidation; ii) clinical assessment defined by worsening or new respiratory symptoms (shortness of breath, cough and dyspnea on exertion) and physical examination findings (wheezing, rhonchi, rales, crackles) iii) New BiPAP requirement or emergent intubation.
Change in oxygen requirement | Starting on admission and continuing for 72 hours
  Measure percentage change in oxygen requirement in each subject in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Imran Naqvi, MD, Principal Investigator — Jewish Hospital of Cincinnati; Nasim Motayar, MD, Principal Investigator — Jewish Hospital of Cincinnati
Locations (1):
- Jewish Hospital of Cincinnati, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided